DigiVis: validation of self-testing visual acuity web-based app to aid ophthalmic telephone consultations during Covid19 lockdown and subsequent social distancing crisis.

## **Clinical Study Protocol**

Protocol Number: DigiVis v0.1

NCT: IRAS ID 196573 Document date: 15<sup>th</sup> July 2020

Study Title: DigiVis: validation of self-testing visual acuity web-based app

to aid ophthalmic telephone consultations during Covid19

lockdown and subsequent social distancing crisis.

Investigational Product: Web-based Visual Acuity software

Protocol Version: Version 0.1

Chief investigator: Miss Louise E Allen MBBS MD MA FRCOphth

Consultant Paediatric Ophthalmologist, Addenbrooke's

Hospital

Investigator's address: Box 41, Ophthalmology Department

Hills Road Cambridge CB2 0QQ

Study Location: Addenbrooke's Hospital, Cambridge (CUHFT)

Telephone: 01223 216700

Study Sponsor: Cambridge University Hospitals NHS Foundation Trust

# 1 Study Synopsis

| software by comparison to current chart-based tests Comparison of VA assessment with DigiVis software to clinic-based VA assessment. Secondary objective (s) Calculation of test-retest variability. Assessment of usability and preference. Study Design Prospective quantifiable comparison study Completed testing on a sufficient number of individuals to give good statistical power. Approximately 250 patients in total Summary of eligibility criteria Patients aged between 5 and 85 due to attend scheduled clinic appointment with vision +0.8logMAR (6/38) or better in their left eye. Patients with access to two appropriate digital devices. Ability to understand English and log on to the website. Active comparator product(s) Clinic VA charts: LogMAR visual acuity chart, SLT childrens' vision chart. Route(s) of administration Visual test Assimum duration of treatment Procedures: Screening & enrolment Procedures: Screening & enrolment Comparators VA test at the scheduled clinic appointment. Telephone enrolment will be undertaken. VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study End of Study Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds | Title of clinical trial | DigiVis: self-testing vision app for telephone consultations |
|---|---|---|
| Medical condition under investigation Purpose of clinical trial Purpose of clinical trial To validate VA self-assessment using DigiVis software by comparison to current chart-based tests Primary objective Comparison of VA assessment. Secondary objective (s) Calculation of test-retest variability. Assessment of usability and preference. Study Design Prospective quantifiable comparison study Completed testing on a sufficient number of individuals to give good statistical power. Sample Size Approximately 250 patients in total Patients aged between 5 and 85 due to attend scheduled clinic appointment with vision +0.8logMAR (6/38) or better in their left eye. Patients with access to two appropriate digital devices. Ability to understand English and log on to the website. Clinic VA charts: LogMAR visual acuity chart, SLT childrens' vision chart. Route(s) of administration Visual test Procedures: Screening & enrolment Procedures: Screening & enrolment Comparators Comparators VA test at the scheduled clinic appointment. The DigiVis self-test VA measurements. Patient preference. Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Scheduled clinic appointment rival Criteria for withdrawal of patients on safety grounds | Sponsor name | Cambridge University Hospitals NHS Trust |
| Purpose of clinical trial Primary objective Primary objective Comparison of VA assessment using DigiVis software by comparison to current chart-based tests Comparison of VA assessment using DigiVis software to clinic-based VA assessment. Secondary objective (s) Calculation of test-retest variability. Assessment of usability and preference. Study Design Prospective quantifiable comparison study Completed testing on a sufficient number of individuals to give good statistical power. Sample Size Approximately 250 patients in total Patients aged between 5 and 85 due to attend scheduled clinic appointment with vision +0.8logMAR (6/38) or better in their left eye. Patients with access to two appropriate digital devices. Ability to understand English and log on to the website. Active comparator product(s) Clinic VA charts: LogMAR visual acuity chart, SLT childrens' vision chart. Visual test Route(s) of administration Visual test Comparators Visual test Procedures: Screening & enrolment Procedures: Screening & enrolment Procedures: Screening & enrolment Procedures: Screening & enrolment Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-test VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study End of Study End of scheduled clinic appointment Tivalic and get usability feedback End of Study End of scheduled clinic appointment Tivalic and get usability feedback End of study End of scheduled clinic appointment Tivalic and get usability feedback End of study Frocedures for safety monitoring during Tival Criteria for withdrawal of patients on Safety grounds | | Visual Acuity (VA) assessment |
| software by comparison to current chart-based tests Comparison of VA assessment with DigiVis software to clinic-based VA assessment. Secondary objective (s) Calculation of test-retest variability. Assessment of usability and preference. Study Design Prospective quantifiable comparison study Completed testing on a sufficient number of individuals to give good statistical power. Approximately 250 patients in total Summary of eligibility criteria Patients aged between 5 and 85 due to attend scheduled clinic appointment with vision +0.8logMAR (6/38) or better in their left eye. Patients with access to two appropriate digital devices. Ability to understand English and log on to the website. Active comparator product(s) Clinic VA charts: LogMAR visual acuity chart, SLT childrens' vision chart. Route(s) of administration Visual test Assimum duration of treatment Procedures: Screening & enrolment Procedures: Screening & enrolment Comparators VA test at the scheduled clinic appointment. Telephone enrolment will be undertaken. VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study End of Study Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds | Purpose of clinical trial | To validate VA self-assessment using DigiVis |
| to clinic-based VA assessment. Secondary objective (s) Calculation of test-retest variability. Assessment of usability and preference. Prospective quantifiable comparison study Study Endpoints Completed testing on a sufficient number of individuals to give good statistical power. Sample Size Approximately 250 patients in total Summary of eligibility criteria Patients aged between 5 and 85 due to attend scheduled clinic appointment with vision +0.8logMAR (6/38) or better in their left eye. Patients with access to two appropriate digital devices. Ability to understand English and log on to the website. Active comparator product(s) Clinic VA charts: LogMAR visual acuity chart, SLT childrens' vision chart. Visual test Maximum duration of treatment Procedures: Screening & enrolment Eligible patients will be identified from electronic patient record prior to a scheduled clinical appointment. Telephone enrolment will be undertaken. VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study End of scheduled clinic appointment n/a Criteria for withdrawal of patients on safety grounds | | |
| Secondary objective (s) Calculation of test-retest variability. Assessment of usability and preference. Prospective quantifiable comparison study Completed testing on a sufficient number of individuals to give good statistical power. Sample Size Approximately 250 patients in total Patients aged between 5 and 85 due to attend scheduled clinic appointment with vision +0.8 logMAR (6/38) or better in their left eye. Patients with access to two appropriate digital devices. Ability to understand English and log on to the website. Clinic VA charts: LogMAR visual acuity chart, SLT childrens' vision chart. Wisual test Procedures: Screening & enrolment Procedures: Screening & enrolment Comparators Comparators Comparators Comparators Intervention period Intervention period End of Study End of Study Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds Comparators Calculation of test-retest variability and preference. Calculation of test-retest variable comparison study Prosedures for safety monitoring during trial Calculation of test-retest variability and preference. Calculation of test-retest variable in cash study Calculation of the sample of safety grounds Calculation of test-retest variability feedback End of Study Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds | Primary objective | Comparison of VA assessment with DigiVis software |
| Assessment of usability and preference. Study Design Prospective quantifiable comparison study Completed testing on a sufficient number of individuals to give good statistical power. Sample Size Approximately 250 patients in total Summary of eligibility criteria Patients aged between 5 and 85 due to attend scheduled clinic appointment with vision +0.8logMAR (6/38) or better in their left eye. Patients with access to two appropriate digital devices. Ability to understand English and log on to the website. Clinic VA charts: LogMAR visual acuity chart, SLT childrens' vision chart. Route(s) of administration Visual test Maximum duration of treatment 2 clinical interventions of 5 minutes each at home Procedures: Screening & enrolment Eligible patients will be identified from electronic patient record prior to a scheduled clinical appointment. Telephone enrolment will be undertaken. VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study End of scheduled clinic appointment n/a Criteria for withdrawal of patients on safety grounds | | to clinic-based VA assessment. |
| Study Design Prospective quantifiable comparison study Study Endpoints Completed testing on a sufficient number of individuals to give good statistical power. Approximately 250 patients in total Summary of eligibility criteria Patients aged between 5 and 85 due to attend scheduled clinic appointment with vision +0.8logMAR (6/38) or better in their left eye. Patients with access to two appropriate digital devices. Ability to understand English and log on to the website. Active comparator product(s) Clinic VA charts: LogMAR visual acuity chart, SLT childrens' vision chart. Route(s) of administration Visual test Maximum duration of treatment 2 clinical interventions of 5 minutes each at home Eligible patients will be identified from electronic patient record prior to a scheduled clinical appointment. Telephone enrolment will be undertaken. Comparators VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study End of scheduled clinic appointment n/a Criteria for withdrawal of patients on safety grounds | Secondary objective (s) | • |
| Study Endpoints Completed testing on a sufficient number of individuals to give good statistical power. Approximately 250 patients in total Patients aged between 5 and 85 due to attend scheduled clinic appointment with vision +0.8logMAR (6/38) or better in their left eye. Patients with access to two appropriate digital devices. Ability to understand English and log on to the website. Active comparator product(s) Clinic Va charts: LogMAR visual acuity chart, SLT childrens' vision chart. Wisual test 2 clinical interventions of 5 minutes each at home Eligible patients will be identified from electronic patient record prior to a scheduled clinical appointment. Telephone enrolment will be undertaken. Comparators Va test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds | | |
| individuals to give good statistical power. Sample Size Approximately 250 patients in total Summary of eligibility criteria Patients aged between 5 and 85 due to attend scheduled clinic appointment with vision +0.8logMAR (6/38) or better in their left eye. Patients with access to two appropriate digital devices. Ability to understand English and log on to the website. Active comparator product(s) Clinic VA charts: LogMAR visual acuity chart, SLT childrens' vision chart. Visual test Maximum duration of treatment 2 clinical interventions of 5 minutes each at home Eligible patients will be identified from electronic patient record prior to a scheduled clinical appointment. Telephone enrolment will be undertaken. VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study End of scheduled clinic appointment n/a Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds | Study Design | Prospective quantifiable comparison study |
| Sample Size Approximately 250 patients in total Patients aged between 5 and 85 due to attend scheduled clinic appointment with vision +0.8logMAR (6/38) or better in their left eye. Patients with access to two appropriate digital devices. Ability to understand English and log on to the website. Active comparator product(s) Clinic VA charts: LogMAR visual acuity chart, SLT childrens' vision chart. Visual test 2 clinical interventions of 5 minutes each at home Eligible patients will be identified from electronic patient record prior to a scheduled clinical appointment. Telephone enrolment will be undertaken. VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds | Study Endpoints | Completed testing on a sufficient number of |
| Summary of eligibility criteria Patients aged between 5 and 85 due to attend scheduled clinic appointment with vision +0.8logMAR (6/38) or better in their left eye. Patients with access to two appropriate digital devices. Ability to understand English and log on to the website. Active comparator product(s) Clinic VA charts: LogMAR visual acuity chart, SLT childrens' vision chart. Visual test Active comparation Visual test Maximum duration of treatment Procedures: Screening & enrolment Comparators Comparators Comparators Comparators Comparators Intervention period Intervention period Intervention period Eligible patients will be identified from electronic patient record prior to a scheduled clinical appointment. Two DigiVis self-test VA measurements. Patient preference. Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study Frocedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds | | individuals to give good statistical power. |
| scheduled clinic appointment with vision +0.8logMAR (6/38) or better in their left eye. Patients with access to two appropriate digital devices. Ability to understand English and log on to the website. Active comparator product(s) Clinic VA charts: LogMAR visual acuity chart, SLT childrens' vision chart. Visual test 2 clinical interventions of 5 minutes each at home Procedures: Screening & enrolment Eligible patients will be identified from electronic patient record prior to a scheduled clinical appointment. Telephone enrolment will be undertaken. VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds | Sample Size | Approximately 250 patients in total |
| +0.8logMAR (6/38) or better in their left eye. Patients with access to two appropriate digital devices. Ability to understand English and log on to the website. Active comparator product(s) Clinic VA charts: LogMAR visual acuity chart, SLT childrens' vision chart. Route(s) of administration Visual test 2 clinical interventions of 5 minutes each at home Procedures: Screening & enrolment Eligible patients will be identified from electronic patient record prior to a scheduled clinical appointment. Telephone enrolment will be undertaken. VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds | Summary of eligibility criteria | Patients aged between 5 and 85 due to attend |
| Patients with access to two appropriate digital devices. Ability to understand English and log on to the website. Active comparator product(s) Clinic VA charts: LogMAR visual acuity chart, SLT childrens' vision chart. Route(s) of administration Maximum duration of treatment Procedures: Screening & enrolment Procedures: Screening & enrolment Comparators Comparators VA test at the scheduled clinic appointment. Telephone enrolment will be undertaken. VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds | | • • |
| devices. Ability to understand English and log on to the website. Active comparator product(s) Clinic VA charts: LogMAR visual acuity chart, SLT childrens' vision chart. Route(s) of administration Maximum duration of treatment Procedures: Screening & enrolment Eligible patients will be identified from electronic patient record prior to a scheduled clinical appointment. Telephone enrolment will be undertaken. VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds | | • • • • |
| Ability to understand English and log on to the website. Active comparator product(s) Clinic VA charts: LogMAR visual acuity chart, SLT childrens' vision chart. Route(s) of administration Maximum duration of treatment Procedures: Screening & enrolment Eligible patients will be identified from electronic patient record prior to a scheduled clinical appointment. Telephone enrolment will be undertaken. Comparators VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds | | |
| website. Active comparator product(s) Clinic VA charts: LogMAR visual acuity chart, SLT childrens' vision chart. Route(s) of administration Maximum duration of treatment Procedures: Screening & enrolment Comparators Comparators Intervention period Intervention period End of Study End of Study Clinic VA charts: LogMAR visual acuity chart, SLT childrens' vision chart. Clinic VA charts: LogMAR visual acuity chart, SLT childrens' vision chart. Visual test 2 clinical interventions of 5 minutes each at home Eligible patients will be identified from electronic patient record prior to a scheduled clinical appointment. Telephone enrolment will be undertaken. VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study End of Study Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds | | |
| Active comparator product(s) Clinic VA charts: LogMAR visual acuity chart, SLT childrens' vision chart. Noute(s) of administration Maximum duration of treatment Procedures: Screening & enrolment Comparators Comparators Comparators Intervention period Intervention period End of Study Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds Cinic VA charts: LogMAR visual acuity chart, SLT childrens' vision chart. Visual test Visual test Visual test 2 clinical interventions of 5 minutes each at home Eligible patients will be identified from electronic patients on sorce scheduled clinical appointment. Telephone enrolment will be undertaken. VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study Procedures for safety monitoring during n/a | | |
| childrens' vision chart. Note(s) of administration Maximum duration of treatment Procedures: Screening & enrolment Eligible patients will be identified from electronic patient record prior to a scheduled clinical appointment. Telephone enrolment will be undertaken. Comparators VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds | | |
| Maximum duration of treatment Procedures: Screening & enrolment Comparators Intervention period Intervention period End of Study End of Study Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds Z clinical interventions of 5 minutes each at home 2 clinical interventions of 5 minutes each at home Eligible patients will be identified from electronic patient record prior to a scheduled clinical appointment. Telephone enrolment will be undertaken. VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of scheduled clinic appointment n/a n/a Telephone enrolment will be identified from electronic patients of vA test at the scheduled clinic appointment n/a | Active comparator product(s) | • |
| Maximum duration of treatment Procedures: Screening & enrolment Eligible patients will be identified from electronic patient record prior to a scheduled clinical appointment. Telephone enrolment will be undertaken. Comparators VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds | | |
| Procedures: Screening & enrolment Eligible patients will be identified from electronic patient record prior to a scheduled clinical appointment. Telephone enrolment will be undertaken. VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study End of Study End of scheduled clinic appointment n/a Criteria for withdrawal of patients on safety grounds The formal prior to a scheduled from electronic patients will be identified from electronic patients will be undertaken. VA test at the scheduled clinic appointment. Two 10 minute phone calls explaining study and the test Two 5 minute patients of VA on the website 10 minute phone calls explaining study and the test Two 5 minute phone calls explaining study and the test Two 5 minute phone calls explaining study and the test | Route(s) of administration | |
| patient record prior to a scheduled clinical appointment. Telephone enrolment will be undertaken. Comparators VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study End of scheduled clinic appointment Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds | Maximum duration of treatment | 2 clinical interventions of 5 minutes each at home |
| appointment. Telephone enrolment will be undertaken. VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study End of scheduled clinic appointment Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds | Procedures: Screening & enrolment | Eligible patients will be identified from electronic |
| Telephone enrolment will be undertaken. VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study End of scheduled clinic appointment n/a Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds | | patient record prior to a scheduled clinical |
| Comparators VA test at the scheduled clinic appointment. Two DigiVis self-test VA measurements. Patient preference. Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study End of scheduled clinic appointment Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds | | • • |
| Two DigiVis self-test VA measurements. Patient preference. Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study End of scheduled clinic appointment Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study n/a n/a | | · |
| Patient preference. Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study End of scheduled clinic appointment Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds Patient preference. Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study n/a n/a | Comparators | • • |
| Intervention period Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study End of scheduled clinic appointment n/a trial Criteria for withdrawal of patients on safety grounds Two 10 minute phone calls explaining study and the test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study n/a | | |
| test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study End of scheduled clinic appointment Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds test Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of scheduled clinic appointment n/a n/a | | • |
| Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study End of scheduled clinic appointment n/a trial Criteria for withdrawal of patients on safety grounds Two 5 minute self-tests of VA on the website 10 minutes conversation to sign the consent form in clinic and get usability feedback In description of the website 10 minutes conversation to sign the consent form in clinic and get usability feedback In description of the website 10 minutes conversation to sign the consent form in clinic and get usability feedback In description of the website 10 minutes conversation to sign the consent form in clinic and get usability feedback In description of the website 10 minutes conversation to sign the consent form in clinic and get usability feedback In description of the website 10 minutes conversation to sign the consent form in clinic and get usability feedback In description of the website 10 minutes conversation to sign the consent form in clinic and get usability feedback In description of the website 10 minutes conversation to sign the consent form in clinic and get usability feedback In description of the website 10 minutes conversation to sign the consent form in clinic and get usability feedback In description of the website 10 minutes conversation to sign the consent form in clinic and get usability feedback In description of the website 10 minutes conversation to sign the consent form in clinic and get usability feedback In description of the website 10 minutes conversation to sign the consent form in clinic and get usability feedback In description of the website 10 minutes conversation of the webs | Intervention period | |
| 10 minutes conversation to sign the consent form in clinic and get usability feedback End of Study End of scheduled clinic appointment n/a trial Criteria for withdrawal of patients on safety grounds 10 minutes conversation to sign the consent form in clinic and get usability feedback End of scheduled clinic appointment n/a n/a | | |
| clinic and get usability feedback End of Study End of scheduled clinic appointment n/a trial Criteria for withdrawal of patients on safety grounds | | |
| End of Study End of scheduled clinic appointment Procedures for safety monitoring during trial Criteria for withdrawal of patients on safety grounds End of scheduled clinic appointment n/a 1/a | | |
| Procedures for safety monitoring during n/a trial Criteria for withdrawal of patients on n/a safety grounds | E. J. Co. J. | |
| trial Criteria for withdrawal of patients on n/a safety grounds | • | • • |
| safety grounds | Procedures for safety monitoring during trial | |
| Regulatory submissions on safety grounds Software marked as CE Class I Medical Device | Criteria for withdrawal of patients on safety grounds | n/a |
| <u> </u> | Regulatory submissions on safety grounds | Software marked as CE Class I Medical Device |

## 2 Introduction

## 2.1 Background

Eye problems like macular degeneration and amblyopia (lazy eye) require regular monitoring to prevent permanent visual impairment. Over 2000 patients a month are seen in CUH eye clinics; concern about Covid-19 infection has led to over 80% of consultations being conducted by telephone with few clinical clues to inform decision making. Patients will face long delays even when routine clinics restart: there is no doubt that some will suffer preventable visual loss.

DigiVis is a web-based vision testing app enabling self-testing of vision at home. Early testing and patient feedback is positive: 80% of children prefer DigiVis to regular testing. We wish to test how accurately the app works for home use, by asking older children and adults to self-test their vision prior to their planned face to face clinic appointment. Once tested, DigiVis will be available free of charge to patients, not only during the Covid-19 crisis, but also to support telephonic consultations in the future.

Visual acuity (VA) is a fundamental measure of vision required for all ophthalmic assessments. It is measured by health professionals using vision charts. DigiVis is a new app which enables self-testing of VA using two wirelessly connected digital devices. By matching letters on a handheld device to those displayed on the second device a distance away, threshold VA can be measured using a staircase algorithm. The distance and scaling of the test is vital to its accuracy and a concept (patent filed by Cambridge Enterprise) in DigiVis enables this without the need for manual distance measurement or an observer.

Early validation using two tablet computers in 150 clinic patients has given positive results, both in testing accuracy and patient feedback. With the current Covid-19 crisis limiting face to face appointments, there is an urgent need for accurate home VA assessment. The DigiVis app has been re-coded for free website delivery for this purpose.

We wish to formally validate DigiVis home testing following CE (class I) marking so that it can be recommended for clinical use. 250 patients will be invited to self-test their VA twice using DigiVis prior to a planned face to face clinic appointment. The test-retest variability and comparison of DigiVis VA to chart based assessment will be compared.

The DigiVis test can be undertaken at <a href="https://www.digivis.org">www.digivis.org</a> with a code name of louiseallen.

#### 2.2 Data from other studies

The DigiVis software app has already undergone initial validation and usability studies in clinic patients, which have resulted in software improvement including a reduction of test time.

A similar study design has been used to assess Peek vision, a smartphone based VA testing app. (1) The difference between DigiVis and Peek app is the automated distance measurement, no requirement for an observer and use of standardised optotype design in the former.

## 2.3 Safety data

The software is CE marked Class1 medical devices and is delivered on a web-site accessed from the patients' own digital devices, no safety issues are foreseen.

## 3 Rationale for Study

Validation of the accuracy of the software package will enable recommendation of its use in conjunction with telephone consultation to inform clinical decision making during and after the lockdown period as social distancing increases the need for virtual consultations.

## 4 Trial objective and purpose

Primary objective: to compare VA assessment of self-testing on the DigiVis website to formal VA measurement using chart-based tests in clinic.

Secondary objective: to assess the repeatability and usability of the software.

## 4.1 Statement of design

This is a prospective quantifiable comparison study.

## 4.2 Study duration

Study duration will be 6 months, aiming to start testing by the 3rd June 2020 and complete testing by 3<sup>rd</sup> February 2021.

## 4.3 Study objectives

#### 4.3.1 Primary research question

Is the visual acuity score measured by home self-testing with DigiVis comparable to current chart-based clinic methods?

#### 4.3.2 Secondary research question

What is the test-retest variation (repeatability) of the DigiVis system? What is the ease of use of the app and what features could be modified to improve usability? Study endpoints

#### 4.3.3 Primary endpoint

Clinical testing will cease once at least 250 individuals have been recruited to enable adequate statistical power using Bland-Altman calculations.

## 4.4 Criteria for Discontinuation

#### 4.4.1 Individual subject

Request of the child or parent to withdraw from study or cease testing.

## 5 Selection and withdrawal of subjects

#### 5.1 Inclusion Criteria

- Age between 5 and 85 years scheduled to have face to face appointment within two weeks
- Previous recorded visual acuity of +0.8logMAR (6/38) or better in the left eye

#### 5.2 Exclusion Criteria

- Individuals with poor conversant English
- Patients with cognitive impairment
- Patients without suitable digital devices or inability to access the internet

## 5.3 Assignment and Randomisation Number

The data regarding VA assessment of the left eye only of individuals will be analysed.

## 5.4 Method of Blinding

The health care assistant or orthoptist undertaking the standard chart-based test will not have knowledge of the DigiVis VA results.

#### 5.5 Emergency Unblinding

Not applicable

#### 5.6 Subject withdrawal criteria

The individual will be withdrawn from the study if it he/she is unable to access the DigiVis website or undertake the test twice.

## 6 Study procedure and assessments

## 6.1 Informed consent

Subjects who fulfil the inclusion criteria will undergo the following consent process:

First telephone call:

The researcher will telephone patients prior to their scheduled face to face clinic appointment for an introductory phone call to explain the study and to determine if any exclusion criteria apply.

If interested in the study at this first contact, the individual will be directed to the website and shown how to access the study information and consent form. The researcher will go over both forms with the potential participant. A convenient time for a follow up call at least 30 minutes after the first will be arranged to allow the patients

to consider participation and discuss with friends and family. They will be informed that non-participation will not affect patient care. Access to the website is possible via a password and no personal information is stored in the web-server.

## Second telephone call:

If the patient wishes to participate in the study they will be asked to read and electronically consent to undertaking the DigiVis test on the website itself. The researcher will then help them undertake the first VA test and will note down the VA values. The participant will be asked to undertake the test themselves a second time before their scheduled clinic appointment and note down, or take a photo of, their VA score.

#### Clinic assessment:

At this appointment, as standard practice, chart-based VA will be assessed by a health care professional (who is masked to the result of the DigiVis scores). A researcher will approach the subject during their visits and the formal study consent form will be signed and the usability feed-back documented.

#### 6.2 Personal data

The personal data recorded for the study will be hospital number and date of birth. Study data will include: DigiVis VA score x 2, chart based VA score, usability score and patient comments.

#### 7 Evaluation of Results

Bland Altman statistical methods and calculation of test-retest variability will be calculated after 100 adults and 150 children have been tested.

## 8 Assessment of Safety

No safety issues are expected during this study because the patients is using their own devices and the clinic element of the study is standard clinical practice.

## 9 Statistics

#### 9.1 Statistical methods to be employed

Bland-Altman statistics similar to those illustrated in the initial validation studies will be used. In addition test-retest variability and quantative comparison of preference and usability will be analysed. Sample size requirements have been calculated using MedCalc based on the results from the initial validation studies (graph 1&2)

## 9.2 Number of Subjects to be enrolled

100 adults 150 children aged 5-16years

#### 9.3 Criteria for the termination of the trial

Website issues, although this is unlikely since the website is already running and tested.

## 9.4 Procedure to account for missing or spurious data

The first DigiVis score will be take down over the telephone at the time of the second call. It is possible that the participant may forget to take the DigiVis a second time or forget to bring the VA score. Where this occurs, the DigiVis test will be repeated in clinic.

#### 9.5 Definition of the end of the trial

Interim data analysis will be undertaken once 100 adults and 150 children have been tested to ensure sufficient statistical power. If insufficient further recruitment may be necessary.

## 10 Direct access to source data / documents

The investigators will permit trial related monitoring, audits, REC review, regulatory inspections.

#### 11 Ethical considerations – none forseen

#### 11.1 Consent

All patients will freely give their informed consent to participate in the study. A patient may decide to withdraw from the study at any time without prejudice to their future care.

Initial electronic consent will be given by parents at the time of their DigiVis testing. Formal written consent will be collected at the time of their clinic attendance.

#### 11.2 Ethical committee review

The study protocol will be submitted to the appropriate ethical review committee with a letters of approval filed in the study file

#### 11.3 Declaration of Helsinki and ICH Good Clinical Practise

The study will be carried out in conformation with the spirit and the letter of the declaration of Helsinki, and in accord with the ICH Good Clinical Practice Guidelines

## 12 Data handling and record keeping

Data with personal information will be kept for analysis 6-12 months following study and subsequently pseudonymised and kept as a file on an NHS hospital computer for a period of 15 years by Miss Allen.

#### 13 Financial and Insurance

This trial has been funded by a combination of Addenbrooke's Charitable Trust and Fight Against Blindness charitable funding. The original coding of DigiVis was enabled by an MRC: Confidence in concepts grant in 2016. The investigators will be working within Cambridge University Hospitals NHS Trust and will be indemnified by the NHS. The VA app will be available free of charge to patients for the foreseeable future.

## 14 Publications policy

Publications arising from the trial will be authored by Miss Allen. If acceptable accuracy and reliability of DigiVis self-assessment is demonstrated, it is likely that the app will be recommended for the use by the Royal College of Ophthalmologists.

## References

1) Bastawrous A, Rono H, Livingstone IA, ey al. The development of a smartphone visual acuity test (Peek acuity) for clinical practice and community based field work. JAMA Ophthalmol. 2015 August;133(8) 930-937